CLINICAL TRIAL: NCT07112313
Title: A Prospective, Observational, Single-Center Study Evaluating Preoperative and Postoperative Changes in the Frontal QRS Axis on Electrocardiogram in Patients Undergoing Total Knee Arthroplasty Under Spinal Anesthesia
Brief Title: Frontal QRS Axis Changes in Patients Undergoing Total Knee Arthroplasty With Spinal Anesthesia (FQRS-TKA)
Acronym: FQRS-TKA
Status: Completed | Type: Observational
Sponsor: Sevim Şenol Karataş (Other)
Responsible Party: Sponsor-Investigator, Sevim Şenol Karataş, Specialist in Anesthesiology, Elazıg Fethi Sekin Sehir Hastanesi
Organization: Elazıg Fethi Sekin Sehir Hastanesi (Other)
Other Study IDs: EFSH-ANES-2025-01
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Spinal Anesthesia; Total Knee Arthroplasty
Keywords: Frontal QRS axis; Spinal anesthesia; Total knee replacement; Electrocardiogram (ECG); Postoperative ECG changes; Regional anesthesia; Orthopedic surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TKA Patients: Patients undergoing elective total knee arthroplasty under spinal anesthesia. Frontal QRS axis will be measured using standard 12-lead ECG preoperatively (within 2 hours before surgery) and postoperatively (within 2 hours after surgery and before mobilization). The study aims to evaluate the change in frontal QRS angle following spinal anesthesia.

SUMMARY:
This prospective, single-center, observational study aims to evaluate changes in the frontal QRS axis on ECG before and after spinal anesthesia in patients undergoing total knee arthroplasty. The primary objective is to determine whether spinal anesthesia causes a significant alteration in the frontal QRS axis. A total of 80 patients will be enrolled, and preoperative and postoperative ECG measurements will be compared using paired t-test or Wilcoxon signed-rank test depending on data distribution.

DETAILED DESCRIPTION:
This study will be conducted in the Department of Anesthesiology and Reanimation at Elazığ Fethi Sekin City Hospital. It is a prospective, observational, and single-center study designed to evaluate the impact of spinal anesthesia on the frontal QRS axis in patients undergoing elective total knee arthroplasty.

The primary endpoint is the difference between preoperative and postoperative frontal QRS axis measurements. ECG recordings will be taken within 2 hours before and after surgery. Frontal QRS axis values will be automatically calculated by the ECG machine and verified manually.

Inclusion criteria include patients aged 45-85 years, ASA class I-III, undergoing spinal anesthesia for elective knee replacement surgery, and able to obtain ECG recordings before and after the procedure. Patients with arrhythmias such as atrial fibrillation or pacemaker dependency, or those requiring postoperative ICU care or general anesthesia conversion will be excluded.

The estimated sample size was calculated using G*Power software. Based on previous studies, a minimum of 34 patients is required to detect a clinically significant change of 10 degrees in QRS axis, with a planned enrollment of 80 patients considering data loss.

Statistical analysis will be conducted using SPSS 26.0. A p-value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 45 and 85 years
* ASA physical status I-III
* Scheduled for elective total knee arthroplasty under spinal anesthesia
* Able to tolerate 12-lead ECG before and within 2 hours after surgery

Exclusion Criteria:

* Known rhythm disorders affecting ECG axis (e.g., heart block, atrial fibrillation, pacemaker)
* Conversion to general anesthesia
* Admission to intensive care unit after surgery
* Missing ECG data
* Communication or mental disorders

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 45-85 years undergoing elective total knee arthroplasty under spinal anesthesia at Elazığ Fethi Sekin City Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Frontal QRS Axis After Spinal Anesthesia | From 2 hours before to 2 hours after surgery
  To evaluate the difference in frontal QRS axis values on the electrocardiogram (ECG) before and after spinal anesthesia in patients undergoing total knee arthroplasty.

CONTACTS AND LOCATIONS:
Overall Officials: Sevim Ş Karataş, MD, Principal Investigator — Elazığ Fethi Sekin City Hospital
Locations (1):
- Elazığ Fethi Sekin City Hospital, Elâzığ, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No